CLINICAL TRIAL: NCT04171414
Title: A Phase III, Open-label, Single-arm, Multiple-dose Study to Evaluate Usability of Subcutaneous Auto-injector of CT-P17 in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Evaluate Usability of Subcutaneous Auto-injector of CT-P17 in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-P17 3.2; 2019-000660-25 (EudraCT Number)
Record Dates: First submitted 2019-09-18; First posted 2019-11-20 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "CT-P17 SC AI (adalimumab)" (Experimental): CT-P17 Subcutaneous(SC) Autoinjector(AI) (adalimumab)
  Interventions: Biological: CT-P17 SC AI (adalimumab)

INTERVENTIONS:
Biological: CT-P17 SC AI (adalimumab) — Subcutaneous Injection of Adalimumab 40mg once every two weeks

SUMMARY:
Clinical trial to evaluate Usability of Subcutaneous Auto-injector of CT-P17 in Patients With Active Rheumatoid Arthritis

DETAILED DESCRIPTION:
CT-P17, containing the active ingredient adalimumab, is a recombinant humanized monoclonal antibody that is being developed as a similar biological medicinal product to Humira. The purpose of this study is to evaluate usability of subcutaneous auto-injector of CT-P17 in patients with moderate to severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 to 70 years, inclusive.
* Patient must be able and willing to self-administer subcutaneous (SC) injections via auto injector (AI).

Exclusion Criteria:

* Patient who has previously received investigational or licensed product; biologic or targeted synthetic disease-modifying antirheumatic drugs for the treatment of rheumatoid arthritis and/or a tumor necrosis factor (TNF) α inhibitor for any purposes.
* Patient who has allergies to any of the excipients of study drug or any other murine and human proteins, or patient with a hypersensitivity to immunoglobulin products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MinJi Ma, Study Chair — Celltrion, Inc.
Locations (1):
- Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- "CT-P17 SC AI (Adalimumab)": The CT-P17 (40mg/0.4mL) was administered every other week (EOW) by subcutaneous (SC) injection via autoinjector (AI) from Week 0 to Week 24 in combination with methotrexate (MTX) and folic acid.
Period: Overall Study
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Started | 62
Completed | 60
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: Years] | 54.0 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 62
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Poland | 62

OUTCOME MEASURES:

1. Primary Outcome: The Usability as Assessed by Patients Rating Using PRE- and POST-Self-Injection Assessment Questionnaire (SIAQ) at Week 4
Description: The usability of CT-P17 Auto Injector is measured by participant using PRE- and POST-Self-injection Assessment Questionnaire (SIAQ) modules. The PRE-SIAQ module is a 7-item questionnaire and the POST-SIAQ module is a 27-item questionnaire that assesses feelings about injections, self-image, self-confidence (regarding self-administration), pain and skin reactions before after injection. Participants rated each item of the SIAQ on a 5-point (or 6-point) semantic Likert-type scal. (each item graded on a 5-point scale). [Scores were transformed to Rate between 0 (worst) to 10 (best)]
Time Frame: Week 4
Population: Usability and Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
scores on a scale
  Feelings about self-injections (PRE) | 8.00 (2.131)
  Feelings about self-injections (POST) | 8.16 (2.036)
  Self-confidence (PRE) | 6.55 (1.859)
  Self-confidence (POST) | 7.07 (1.616)
  Self-image (POST) | 8.39 (2.079)
  Pain and skin reactions during or after the injection (POST) | 9.59 (0.968)
  Ease of use of the self-injection device (POST) | 8.70 (1.457)
  Satisfaction with self-injection (PRE) | 8.27 (1.669)
  Satisfaction with self-injection (POST) | 8.23 (1.191)

2. Secondary Outcome: Patient's Rating of PRE- and POST-SIAQ at Weeks 0, 2, and 24
Time Frame: Week 0
Population: Usability and Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
scores on a scale
  Feelings about self-injections (PRE) | 7.39 (2.437)
  Feelings about self-injections (POST) | 8.04 (2.086)
  Self-confidence (PRE) | 5.22 (2.272)
  Self-confidence (POST) | 6.18 (2.518)
  Self-image (POST) | 8.35 (2.306)
  Pain and skin reactions during or after the injection (POST) | 9.48 (1.152)
  Ease of use of the self-injection device (POST) | 8.40 (1.531)
  Satisfaction with self-injection (PRE) | 6.15 (1.682)
  Satisfaction with self-injection (POST) | 8.00 (1.250)

3. Secondary Outcome: Observer's Rating of Successful Self-injection Using Self-injection Assessment Checklist at Weeks 0, 2, 4, and 24
Time Frame: Week 0,2,4,24
Population: Usability and Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
Participants
  Week 0, Successful Self-Injection | 62
  Week 0, Overall Successful Self-Injection | 62
  Week 2, Successful Self-Injection | 62
  Week 2, Overall Successful Self-Injection | 62
  Week 4, Successful Self-Injection | 62
  Week 4, Overall Successful Self-Injection | 62
  Week 24, Successful Self-Injection | 60
  Week 24, Overall Successful Self-Injection | 60

4. Secondary Outcome: Mean for Actual Values and Change From Baseline in DAS28 (CRP and ESR)
Description: DAS28 (CRP) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(CRP+1) + 0.014 X GH on VAS + 0.96. DAS28 (CRP) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
  DAS28 (ESR) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(ESR) + 0.014 X GH on VAS. DAS28 (ESR) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
  Abbreviation: CRP, C-reactive protein; DAS28, Disease Activity Score using 28 joint counts; ESR, Erythrocyte sedimentation rate
Time Frame: Week 8,16,24
Population: ITT population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
scores on a scale
  CRP, Baseline | 5.248 (0.8415)
  CRP, Week 8, Change from baseline | -2.560 (1.1223)
  CRP, Week 16, Change from baseline | -2.795 (1.2381)
  CRP, Week 24, Change from baseline | -3.111 (1.1109)
  ESR, Baseline | 6.190 (0.7360)
  ESR, Week 8, Change from baseline | -3.287 (1.3525)
  ESR, Week 16, Change from baseline | -3.495 (1.4695)
  ESR, Week 24, Change from baseline | -3.799 (1.4287)

5. Secondary Outcome: Patient's Rating of PRE- and POST-SIAQ at Weeks 0, 2, and 24
Time Frame: Week 2
Population: Usability and Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
scores on a scale
  Feelings about self-injections (PRE) | 7.93 (2.175)
  Feelings about self-injections (POST) | 8.08 (2.110)
  Self-confidence (PRE) | 6.61 (2.007)
  Self-confidence (POST) | 6.67 (1.811)
  Self-image (POST) | 8.27 (2.245)
  Pain and skin reactions during or after the injection (POST) | 9.64 (0.693)
  Ease of use of the self-injection device (POST) | 8.34 (1.698)
  Satisfaction with self-injection (PRE) | 7.78 (2.128)
  Satisfaction with self-injection (POST) | 8.16 (1.177)

6. Secondary Outcome: Patient's Rating of PRE- and POST-SIAQ at Weeks 0, 2, and 24
Time Frame: Week 24
Population: Usability and Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | "CT-P17 SC AI (Adalimumab)"
Number analyzed (Participants) | 62
scores on a scale
  Feelings about self-injections (PRE) | 8.88 (2.034)
  Feelings about self-injections (POST) | 8.97 (1.888)
  Self-confidence (PRE) | 7.21 (1.556)
  Self-confidence (POST) | 7.44 (1.840)
  Self-image (POST) | 9.04 (1.533)
  Pain and skin reactions during or after the injection (POST) | 9.60 (0.841)
  Ease of use of the self-injection device (POST) | 9.35 (1.057)
  Satisfaction with self-injection (PRE) | 8.83 (1.868)
  Satisfaction with self-injection (POST) | 8.95 (1.023)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the patient signed the ICF until EOS/ED visit. (up to week 28, including 4 weeks of follow-up period)
Arm/Group | "CT-P17 SC AI (Adalimumab)"
All-Cause Mortality (participants affected / at risk) | 1/62
Serious Adverse Events (participants affected / at risk) | 3/62
Other Adverse Events (participants affected / at risk) | 20/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "CT-P17 SC AI (Adalimumab)" (N=62)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (62)
Tooth infection (Infections and infestations) | 1 (62)
Cervical polyp (Reproductive system and breast disorders) | 1 (62)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "CT-P17 SC AI (Adalimumab)" (N=62)
Upper respiratory tract infection (Infections and infestations) | 13 (62)
Urinary tract infection (Infections and infestations) | 3 (62)
Diarrhoea (Gastrointestinal disorders) | 2 (62)
Headache (Nervous system disorders) | 2 (62)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (62)
Influenza like illness (General disorders) | 2 (62)
Injection site reaction (General disorders) | 2 (62)
Nasopharyngitis (Infections and infestations) | 2 (62)
Pharyngitis (Infections and infestations) | 2 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04171414/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04171414/SAP_001.pdf